CLINICAL TRIAL: NCT04164420
Title: Oral Neuromuscular Training in Stroke Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004:M-435
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Dysphagia
Keywords: Stroke; Dysphagia; Treatment; Intervention
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for five weeks. To either oral neuromuscular training and orofacial sensory-vibration stimulation or to only orofacial sensory-vibration stimulation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral neuromuscular training and orofacial sensory-vibration (Experimental): Intensive training with oral neuromuscular training and orofacial sensory-vibration stimulation for 5 weeks. The oral neuromuscular training is performed three times per session, and three times daily before eating. Regarding the orofacial sensory-vibration stimulation, the instructions is given on how to stimulate the buccinator mechanism, lips, external floor, and the tongue three times daily before a meal by using a toothbrush.
  Interventions: Behavioral: Oral neuromuscular training and orofacial sensory-vibration
- Orofacial sensory-vibration stimulation (Active Comparator): Orofacial sensory-vibration stimulation by using an electrical toothbrush for five weeks. Instructions is given on how to stimulate the buccinator mechanism, lips, external floor, and the tongue three times daily before a meal.
  Interventions: Behavioral: Orofacial sensory-vibration stimulation

INTERVENTIONS:
Behavioral: Oral neuromuscular training and orofacial sensory-vibration — Oral neuromuscular training is performed by using an oral device. The device is placed pre-dentally behind closed lips, and the participant is sitting in an up-right position. The participant is the instructed to hold the device against a gradually-increasing horizontal pulling force for 5-10 s, whilst trying to resist the force by tightening the lips and pressing the head backward against a head rest.
  Arms: Oral neuromuscular training and orofacial sensory-vibration
Behavioral: Orofacial sensory-vibration stimulation — All participants in the control group is given orofacial sensory-vibration stimulation by using an electrical toothbrush. Instructions is given on how to stimulate the buccinator mechanism, lips, external floor, and the tongue three times daily before a meal.
  Arms: Orofacial sensory-vibration stimulation

SUMMARY:
This study aims to explore if oral neuromuscular training is superior to orofacial sensory-vibration stimulation in patients with oropharyngeal dysphagia.

Four weeks after stroke onset, patients with oropharyngeal dysphagia and pathological swallowing according to the timed water swallow test (TWST) will be randomized 1:1 into a 5-week oral neuromuscular training with an oral device in addition to orofacial sensory-vibration stimulation with an electrical toothbrush (intervention group) or orofacial sensory-vibration stimulation only (control group). The participants will be examined with a TWST, lip force test, and videofluoroscopy (VFS) of oropharyngeal swallowing before (baseline), after 5-weeks training (end-of-training) and at a 12-18 months follow-up. The primary endpoint is changes in TWST at the end-of-training compared with baseline, and at late follow-up based on intention-to-treat analyses. The secondary endpoints are the corresponding changes in lip force and aspiration frequency at VFS.

DETAILED DESCRIPTION:
This study aims to explore if oral neuromuscular training is superior to orofacial sensory-vibration stimulation in patients with oropharyngeal dysphagia.

Study design: This 2-center study is an intension-to-treat prospective randomized open-label trial with blinded evaluators (PROBE) design. Evaluations are made at baseline, at end of training, and at late follow-up after a period without training to investigate if any lasting positive training effect was present.

Inclusion criteria: First-ever stroke and a pathological timed water swallow test (TWST) at four to five weeks after stroke onset.

Exclusion criteria: Inability to cooperate, percutaneous endoscopic gastrostomy (PEG), neurological diseases other than stroke, known history of dysphagia, prominent horizontal overbite, hypersensitivity to the acrylate in the oral device.

Study procedure: Four weeks after stroke onset, patients with oropharyngeal dysphagia and pathological swallowing according to the timed water swallow test (TWST) will be randomized 1:1 into a 5-week oral neuromuscular training with an oral device in addition to orofacial sensory-vibration stimulation with an electrical toothbrush (intervention group) or orofacial sensory-vibration stimulation only (control group). The participants will be examined with a TWST, lip force test, and videofluoroscopy (VFS) of oropharyngeal swallowing before (baseline), after 5-weeks training (end-of-training) and at a 12-18 months follow-up. The primary endpoint is changes in TWST at the end-of-training compared with baseline, and at late follow-up based on intention-to-treat analyses. The secondary endpoints are the corresponding changes in lip force and aspiration frequency at VFS.

Sample size: In order to detect a critical change with a power of 80 %, a sample size of 44 patients (22 in the intervention group and 22 in the control group) that fulfilled the study protocol was required for a type I error of 5 %.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke and,
* Pathological timed water swallow test (TWST) at four to five weeks after stroke onset.

Exclusion Criteria:

* Inability to cooperate
* Percutaneous endoscopic gastrostomy (PEG)
* Neurological diseases other than stroke
* Known history of dysphagia
* Prominent horizontal overbite
* Hypersensitivity to the acrylate in the oral device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Swallowing ability | Baseline, after end-of-treatment (5 weeks), and at 12-18 months follow-up
  Change in swallowing function measured by the timed water swallow test

SECONDARY OUTCOMES:
Lip-force (LF) | Baseline, after end-of-treatment (5 weeks), and at 12-18 months follow-up
  Change in lip-force measured in newtons (N) with the Lip Force Meter LF100.
Swallowing function | Baseline, after end-of-treatment (5 weeks), and at 12-18 months follow-up
  Change in structural and functional swallowing ability measured by Videofluoroscopy (VFS) by using the penetration-aspiration scale by Rosenbek. The scale ranges from 0 (normal swallowing function) to 8 (aspiration without sufficient coughing/clearance)

CONTACTS AND LOCATIONS:
Overall Officials: Per Wester, Professor, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Hagglund P, Hagg M, Levring Jaghagen E, Larsson B, Wester P. Oral neuromuscular training in patients with dysphagia after stroke: a prospective, randomized, open-label study with blinded evaluators. BMC Neurol. 2020 Nov 7;20(1):405. doi: 10.1186/s12883-020-01980-1. PMID 33158423